CLINICAL TRIAL: NCT06652477
Title: Evaluation of Desmoglein-3 Autoantibodies in the Tissues of Atrophic/Bullous Erosive Oral Lichen Planus and Correlation with Disease Severity
Brief Title: Evaluation of Desmoglein-3 Autoantibodies in the Tissues of Oral Lichen Planus and Correlation with Disease Severity
Status: Not yet recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Doaa abdelwadood mohamed ibrahim essa, Master's degree student, Faculty of Dentistry, Ain Shams University., Ain Shams University
Other Study IDs: Dsg3 in oral lichen planus
Record Dates: First submitted 2024-10-18; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Lichen Planus, Oral
MeSH Terms: conditions — Lichen Planus, Oral

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- groupe A: patients with atrophic boullos erosive oral lichen planus
  Interventions: Diagnostic Test: ELISA
- groupe B: healthy patients
  Interventions: Diagnostic Test: ELISA

INTERVENTIONS:
Diagnostic Test: ELISA — ElISA kit to detect autoantibodies against desmoglein 3 in tissues of oral lichen planus lesions

SUMMARY:
1. evaluate the level of Dsg3 autoantibodies in tissue biopsy of Atrophic/Bullous Erosive (A/BE) OLP (Primary Objective).
2. correlate the severity of the disease with the level of tissue Dsg3 autoantibodies (Secondary Objective).

DETAILED DESCRIPTION:
Oral lichen planus (OLP), a chronic disease and one of the most common dermatoses of the oral mucosa, is characterized by white streaks in a lacelike pattern on the tongue and/or buccal mucosa. The disease is also accompanied by chronic inflammation, the degree of which, correlates with the intensity of the symptoms.

OLP occurs more frequently than the cutaneous form and tends to be more persistent and more resistant to treatment. It aﬀects one to two percent of the general adult population, with a higher prevalence in the female gender, and occurs predominantly in adults over 40, although younger adults and children may be aﬀected .

The most common site of oral involvement is the buccal mucosa followed by the tongue and gingiva, but any site of the oral mucosa can be affected. Clinically, OLP is classified as reticular, atrophic, erosive, plaque-type, and bullous. The reticular pattern is the most common form. It is generally asymptomatic and requires no treatment. In contrast, atrophic-erosive forms usually manifest as erythematous, ulcerative lesions associated with symptoms, fluctuating from mild burning sensation to severe pain, interfering with eating and speaking .

Furthermore, OLP is considered a potentially malignant disorder with a transformation rate of about 1.09%, with greater risk among those with atrophic-erosive forms.

The etiology and pathogenesis of OLP are not completely understood. Several factors have been implicated in the etiology and several hypotheses have been proposed for its pathogenesis.

It is believed that OLP represents an abnormal immune reaction in which keratinocytes are recognized as an antigen, secondary to changes in the antigenicity of the cell surface. This elicits an immune response characterized by invasion of inflammatory cells into the subepithelial layer of connective tissue with degeneration of the epithelium of the basement membrane However, the antigen or antigens triggering factors have not been identified.

Many controversies exist about the pathogenesis of OLP. A large body of evidence supports the role of immune dysregulation in the pathogenesis. The various mechanisms hypothesized to be involved in immunopathogenesis include humoral immunity, antigen-speciﬁc cell-mediated immune response, non-speciﬁc mechanisms, and autoimmune response.

Humoral immunity has been reported to play a role in the pathogenesis of OLP in addition to the presence of immunoglobulins, fibrinogen, and C3 complement in the basement membrane at the lesional and perilesional tissue Furthermore, concentrations of salivary IgG and IgA subclasses may be changed .

Antigen-speciﬁc mechanisms in OLP include antigen presentation by basal keratinocytes, followed by antigen-speciﬁc keratinocyte killing by CD8+ cytotoxic T-cells.

Non-speciﬁc mechanisms include mast cell degranulation and matrix metalloproteinase activation in OLP lesions. These mechanisms may combine to cause T-cell accumulation in the superﬁcial lamina propria, basement membrane disruption, intra-epithelial T-cell migration, and keratinocyte apoptosis .

The possibility of the presence of circulating antibodies was previously indicated against desmoglein 3 (Dsg3) in patients with OLP.

Desmogleins (Dsgs) are the main components of cellular coherence in the epidermis and mucosal surfaces. They are consisting of (Dsg1), (Dsg2), (Dsg3), and (Dsg4). Dsg3 antigen is expressed in the basement membrane zone of the epidermis keeping the cells from detachment.

Dsgs are the victims of autoantibody reaction in some autoimmune bullous diseases such as pemphigus vulgaris and bullous pemphigoid causing disruption of desmosomes and consequent acantholysis.

In 2006, Lukac et al. demonstrated significantly higher concentrations of circulating autoantibodies against Dsg3 among erosive OLP patients and in patients with reticular OLP .

In a recent study including 100 OLP patients, 65% of the patients showed the presence of at least one type of autoantibodies in their serum. Dsg3 autoantibody was positive in 16% of the patients .

Furthermore, Saad et al, in 2018, showed increased levels of Dsg3 autoantibodies in the serum of patients with erosive OLP at baseline and after the use of topical Tacrolimus 0.1%. The results revealed a statistically significant decrease in the level of Dsg3 autoantibodies during the follow-up period.

In 2022, El-Rifaie et al detected that the level of Dsg3 autoantibodies in the serum of OLP patients was significantly higher as compared to normal control persons.

However, it is difficult to infer whether the anti-Dsg3 autoantibodies in lichen planus are of primary pathogenic significance or are a result of epitope spreading which is known to occur in autoimmune diseases. These autoantibodies may be increased as an etiologic agent in OLP or due to inflammatory damage to basal keratinocytes. This damage releases the Dsg3 proteins which act as auto-antigens for autoantibodies formation in the circulatory blood .

All the studies were concerned with detecting Dsg3 autoantibodies level in the serum of OLP patients. Unfortunately, such results do not prove the source of Dsg3 autoantibodies to be the OLP lesions. Thus, the present study will be carried out to detect the level of Dsg3 autoantibodies in tissues affected by atrophic/bullous erosive OLP trying to elucidate the actual role of Dsg3 autoantibodies in the etiopathogenesis of OLP.

ELIGIBILITY:
Inclusion Criteria:

* 1. Males or females suffering from A/BE OLP. 2. Proven diagnosis of oral lichen planus based on criteria of WHO (World Health Organization) which is a clinical criteria, clinically proven painful A/BE form of OLP confirmed by the presence of red or erythematous changes, or shallow ulcerations with fine lacy lines at the periphery of the lesion accentuated by stretching and not eliminated by rubbing (Wickham's striae).

Histopathologically, proven Bullous/erosive or reticular forms of OLP confirmed by the presence of accepted histopathological criteria for lichen planus; basal cell liquefaction, band-like lymphocytic infiltrate at the epithelial-stromal junction with degeneration of basal cell region.

Exclusion Criteria:

* 1. History of drug-induced lichenoid lesions. 2. Presence of systemic conditions such as serious active or recurrent infections, malignancy, diabetes mellitus, hypertension, or significant heart, liver, or renal diseases.

  3. Pregnancy or breastfeeding. 4. History of previous treatments potentially effective on OLP such as antimalarial agents, retinoids, corticosteroids, or immunosuppressive drugs from less than 2 weeks for topical medications, and 4 weeks for systemic medications prior to starting the study.

  5. Loss of pliability or flexibility in the tissues involved by the oral lesions of lichen planus.

  6. Histological signs of epithelial dysplasia or lichenoid lesions within the biopsied sites.

  7. Patient refuses to participate in the study. 8. Vulnerable groups (handicapped, orphans, and prisoners).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study is designed to be a case-control study with a convenience sample size of (20) Participants, will be recruited from the Out-patient Clinic of Oral Medicine, Periodontology and Oral Diagnosis Department, Faculty of Dentistry Ain-Shams University or referred to it.
  The participants who will meet the eligibility criteria will be enrolled into one of the following groups • Group A: (10) participants suffering from oral lichen planus (atrophic bullous erosive pattern).
  • Group B: (10) healthy control participants. Tissue samples from the control group will be obtained from excess tissue from periodontal surgeries, mainly crown lengthening surgeries and implant placement surgeries (avoiding any periodontally affected teeth)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-11-05 (Estimated); Primary Completion 2024-12-05 (Estimated); Study Completion 2024-12-05 (Estimated)

PRIMARY OUTCOMES:
evaluate the level of Dsg3 autoantibodies in tissue biopsy of Atrophic/Bullous Erosive oral lichen planus | baseline
  valuate the level of Dsg3 autoantibodies by ELISA kit trying to elucidate the actual role of Dsg3 autoantibodies in the etiopathogenesis of OLP.

SECONDARY OUTCOMES:
correlate the severity of the disease with the level of tissue Dsg3 autoantibodies | baseline
  we will evaluate the disease severity by Clinical scoring system and correlate it with the level of autoantibodies

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Amr, Principal Investigator — ain shamsh university; yasmeen foaad, Study Director — ain shamsh university

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roopashree MR, Gondhalekar RV, Shashikanth MC, George J, Thippeswamy SH, Shukla A. Pathogenesis of oral lichen planus--a review. J Oral Pathol Med. 2010 Nov;39(10):729-34. doi: 10.1111/j.1600-0714.2010.00946.x. Epub 2010 Oct 4. PMID 20923445
- [Background] Vahide L, Zahra H, Forugh G, Nazi S. Autoantibodies to desmogleins 1 and 3 in patients with lichen planus. Arch Dermatol Res. 2017 Sep;309(7):579-583. doi: 10.1007/s00403-017-1756-x. Epub 2017 Jul 3. PMID 28674915
- [Background] Lukac J, Brozovic S, Vucicevic-Boras V, Mravak-Stipetic M, Malenica B, Kusic Z. Serum autoantibodies to desmogleins 1 and 3 in patients with oral lichen planus. Croat Med J. 2006 Feb;47(1):53-8. PMID 16489697
- [Derived] Abdelwadood D, Fouad YA, El-Khazragy N, Amr AEH. Desmoglein-3 autoantibodies in tissues of oral lichen planus patients and its correlation with disease severity: case-control study. BMC Oral Health. 2025 Jun 6;25(1):930. doi: 10.1186/s12903-025-06303-9. PMID 40481453